CLINICAL TRIAL: NCT00081809
Title: A Phase II Trial of Active Specific Immunotherapy in Patients With Indolent Lymphoma Using Autologous Lymphoma-Derived Heat Shock Protein-Peptide Complex (HSPPC-96)
Brief Title: A Safety and Effectiveness Study of Vaccine Therapy in Patients With Indolent Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-100-09; MDACC Protocol ID99-354
Record Dates: First submitted 2004-04-20; First posted 2004-04-23 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma, Follicular; Lymphoma, Small Lymphocytic
Keywords: non-Hodgkin's lymphoma; Brill-Symmers Disease; Follicular Lymphoma; Lymphoma, Giant Follicular; Lymphoma, Nodular; Follicular Lymphoma, Giant; Giant Follicular Lymphoma; Lymphocytic Lymphoma, Diffuse, Well-Differentiated; Lymphocytic Lymphoma, Well-Differentiated; Lymphoma, Lymphocytic, Diffuse, Well-Differentiated; Lymphoma, Lymphocytic, Well-Differentiated; Lymphoma, Lymphoplasmacytoid, CLL; Lymphoma, Small Lymphocytic, Plasmacytoid; Lymphoplasmacytoid Lymphoma, CLL; Diffuse Well-Differentiated Lymphocytic Lymphoma; Lymphocytic Lymphoma, Diffuse, Well Differentiated; Lymphocytic Lymphoma, Well Differentiated; Lymphoma, Lymphocytic, Diffuse, Well Differentiated; Lymphoma, Lymphocytic, Well Differentiated; Lymphoma, Mucosa-Associated Lymphoid Tissue; MALT Lymphoma; Lymphoma of Mucosa-Associated Lymphoid Tissue; Mucosa-Associated Lymphoid Tissue Lymphoma; Monocytoid B-cell lymphoma; Waldenstrom's macroglobulinemia; Marginal zone lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia

INTERVENTIONS:
Drug: autologous human tumor-derived HSPPC-96

SUMMARY:
Primary Objectives:

* To document the efficacy of treatment with autologous lymphoma-derived HSPPC-96 of selected patients with indolent lymphoma. The efficacy endpoints are:
* the rate of complete and partial responses
* the time to progression.

Secondary Objectives:

* To evaluate the safety and tolerability of autologous tumor-derived heat-shock protein peptide complex (HSPPC-96) administered intradermally once weekly for four consecutive weeks, followed by HSPPC-96 administered once every two weeks.
* To evaluate the feasibility of autologous HSPPC-96 preparation from lymphoma specimens.
* To assess approximately the composition of the tissue source of the autologous HSPPC-96 for each patient.
* To study the effect of autologous lymphoma-derived HSPPC-96 vaccine therapy on the expression of Fas ligand and TRAIL death proteins in peripheral blood lymphocytes of patients with indolent lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated or newly diagnosed follicular center cell grade I or grade II lymphoma, small lymphocytic lymphoma, MALT lymphoma, monocytoid B-cell lymphoma, Waldenstrom's macroglobulinemia, or marginal zone lymphoma with bidimensionally measurable disease;
* Part of the resected specimen must undergo routine pathologic examination to confirm the diagnosis of lymphoma. The remaining tissue must be used for the preparation of autologous HSPPC-96;
* Autologous HSPPC-96 vaccine must be successfully prepared and provided by the sponsor;
* A minimum of 2 grams of non-necrotic, resectable malignant lymphoma for HSPPC-96 preparation;
* Bidimensionally measurable disease in at least one location other than the resected lymphoid tissue;
* Life expectancy of at least 16 weeks;
* Zubrod performance status of less then or equal to 2;
* Adequate bone marrow function;
* Adequate hepatic function;
* Adequate renal function;
* Signed written informed consent;
* Patients of child-bearing potential must practice contraception, which is adequate in the opinion of the Principal Investigator;
* Patients of child-bearing potential must have a negative serum pregnancy test prior to entry into the study and must not be lactating;
* Patients must be willing to be followed at the M. D. Anderson Cancer Center during the course of treatment and follow-up;
* Electrocardiogram if none performed in the prior six months;
* Patients must have no chemotherapy, immunotherapy, radiotherapy, or experimental anti-cancer therapy within six weeks prior to starting autologous HSPPC-96 administration;
* Patients must have fully recovered from prior anti-cancer therapy;
* Tumor measurements and staging no more than 4 weeks prior to receiving the first dose of autologous HSPPC-96.

Exclusion Criteria:

* Patients with active or prior history of central nervous system lymphoma;
* Patients with serious intercurrent medical illnesses, requiring hospitalization;
* Patients with a history of primary or secondary immunodeficiency (other than related to the malignant lymphoma because treatment is dependent on functional immune system) or patients taking immunosuppressive drugs such as systemic corticosteroids;
* Women who are pregnant or lactating;
* Patients participating in another clinical trial;
* Patients receiving growth factors of any kind, including G-CSF, GM-CSF, or Epogen;
* Patients with bulky disease, defined as greater than 10 cm in diameter;
* Patients with positive HIV antibody;
* Patients with more than 4 previous treatment regimens will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2000-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States